CLINICAL TRIAL: NCT06619470
Title: Brain Wave Entrainment Using Alpha Frequency Binaural Beats on Adolescent Swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0303388
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2016-11

CONDITIONS: Athletes
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- binaural beat group (Experimental): Binaural Beats added to music and mental training sessions
  Interventions: Other: binaural beats
- music therapy group (Sham Comparator): music and mental training sessions
  Interventions: Other: binaural beats

INTERVENTIONS:
Other: binaural beats — binaural beats
  Other Names: music therapy

SUMMARY:
Relaxation techniques and binaural beats added to music have a positive effect on athletic performance of swimmers than music therapy and mental training alone

DETAILED DESCRIPTION:
EEG measurement after Relaxation techniques and binaural beats added to music have been employed showed a positive effect on the athletic performance of swimmers when BB have been added to music therapy and mental training

ELIGIBILITY:
Inclusion Criteria:

- adolescent swimmer

Exclusion Criteria:

-

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
reaction time | 6 weeks
  time from stimulus application till response
EEG frequency | 6 weeks
  Brain wave frequency

IPD SHARING:
Plan to Share IPD: No